CLINICAL TRIAL: NCT03020381
Title: Gait as Predictor of Cognitive Decline, Dementia, and Risk of Falls in MCI. A Cohort Study
Brief Title: Gait as Predictor of Dementia and Falls. The Gait and Brain Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Manuel Montero Odasso (Other)
Responsible Party: Sponsor-Investigator, Manuel Montero Odasso, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Other Study IDs: 17200
Record Dates: First submitted 2017-01-06; First posted 2017-01-13 (Estimated); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Gait Apraxia; Mild Cognitive Impairment; Subjective Cognitive Impairment; Cerebral Atrophy; Alzheimer Disease; Dementia
MeSH Terms: conditions — Gait Apraxia; Cognitive Dysfunction; Alzheimer Disease; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — APOEε4 carrier status will be determined by PCR of genomic DNA extracted from anticoagulated blood. Carrier status is determined by dichotomizing into ε4- (ε2/ε3 heterozygote or ε2/ε3 homozygote) and ε4+ (ε4 homozygote or ε4 heterozygote) for consistency with previous studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cognitively Normal (Control Group): Participants aged 60 and older, with absence of Dementia (by DSM IV and DSM V) criteria. Normal age-, sex-, and education-adjusted performance on standardized cognitive tests, which are used to classify mild cognitive impairment (MCI) or prodromal AD.
- Subjective Cognitive Impairment (SCI): Participants aged 60 and older, with absence of Dementia (by DSM IV and DSM V) criteria. Normal age-, sex-, and education-adjusted performance on standardized cognitive tests, which are used to classify mild cognitive impairment (MCI) or prodromal AD. Self-experienced persistent decline in cognitive capacity in comparison with a previously normal status and unrelated to an acute event. Answering "yes" to both of the following questions: "Do you feel like your memory or thinking is becoming worse?" and "Does this concern you?"
- Mild Cognitive Impairment (MCI): Participants aged 60 and older that have self-experienced persistent decline in cognitive capacity and unrelated to an acute event. MCI is operationalized following Peterson's criteria as: i) presence of subjective memory complaints from the patient and family; ii) objective memory impairment in cognitive tests (below 1.5 SD on standardized cognitive tests adjusted by age, sex, and education-); iii) preserved activities of daily living (assessed using the Lawton-Brody scale); iv) absence of clinical dementia established using DSM-IV-TR (from 2007 to 2013) and DSM V (from 2014 and onwards)

SUMMARY:
Motor slowing and cognitive slowing are more prevalent as we age. Importantly, the presence of both in an older person increases their risk of having dementia by ten times. Currently, there are no clinically meaningful predictors of progression to dementia in people with mild cognitive impairment (MCI). The main hypothesis is that subtle variations in gait while performing a simple cognitive task is a reliable, easy to perform, and feasible methodology to detect those older adults at higher risk of progression to dementia and also, at higher risk of further mobility decline and falls.

Rationale. The Canadian population is aging. According to recent estimates, the proportion of the population aged 65 and older will increase rapidly from 13% in 2005 to 25% by 2031. This increase in proportion is accompanied by a considerable amount of disability and subsequent dependency which has major effects on both the quality of life of older adults and their caregivers, and on the Canadian health care system. An important goal of geriatric medicine is to reduce the gap between life expectancy and disability-free life expectancy by reducing disability and dependency in the later years of life. A substantial portion of this disability stems from two major geriatric syndromes: cognitive impairment and mobility limitation. The ultimate manifestations of these syndromes are dementia and falls. Interestingly, these manifestations often coexist in elderly people: falling is a common geriatric syndrome affecting about a third of older adults each year, and dementia affects about a third of Canadians aged 80 and over. Together, dementia and falls are responsible for much of the discomfort, disability, and health care utilization in older adults and each will become more prevalent as older Canadians are expected to number approximately $9 million by 2031. The combined direct cost of dementia and falls for the Canadian Health System is over $4.9 billion per year.

Establishing reliable and easy to obtain predictors to accurately identify MCI patients at highest risk of progressing to dementia is essential first, to determine who will benefit from additional and/or invasive testing and second, to implement preventative strategies, including cognitive training, physical exercises, and aggressive vascular risk factors correction to delay progression. Even a modest one-year delay in dementia incidence could save Canada $109 billion over 30 years.

DETAILED DESCRIPTION:
This longitudinal cohort study started in 2007 and is aiming to assess 600 older persons (60 y/o to 85 y/o) at risk of development cognitive impairment and dementia, during a 25 year of follow-up, since we expanded the study to recruit more participants, which was approved by our Institutional Research Board. The follow-up period was selected in order to cover the potential progression to dementia of at least two-third of the participants. From 2007 to 2023, for the first five years of follow up, assessments were conducted at baseline and every 6 months; since 2023, this was changed by which assessments are being conducted every 12-months along with performing a virtual assessment of outcomes only, every 6-months. After the visit at 60 months, participants will then be followed once a year for 20 years. The six months period between assessments during the first 5 years was selected since it is the minimum time required for detecting significant changes between assessments in cognitive measurements and for avoiding testing learning effects. If changes are not noted within the first five years, then the annual follow-up period will provide sufficient time periods to detect significant changes in cognition, gait, and balance measures.

Blood test for genotyping (ApoE4 carrier) is being performed only at baseline assessments. Cognitive, gait and balance assessments are being performed in all 12-month follow-up visits. From 2010 to 2021, 3Tesla Magnetic Resonance Imaging (structural and functional -resting state-) and MRI spectroscopy are being performed at four different time points: at baseline, month 18 and month 36, and month 60, following the Canadian Dementia Imaging protocol (http://www.cdip-pcid.ca.). Since 2021, the 18-month MRI timepoint changed to be performed at 12-month visit to align MRI timepoints with blood draw, which allows analysis of MRI and biomarker comparisons over time. For the 20-month Follow-Up period, MRI was performed at Year-2, Year-5 and Year-7 until 2018. Since 2018, the 20-Year Follow-Up MRI timepoints changed to Year-3, Year-5, Year-7 and Year-10. Blood and brain imaging were added after the second wave of the study, in 2010.

ELIGIBILITY:
General Inclusion Criteria:

* Absence of Dementia (DSM IV-TR or DSM V criteria)
* Aged 60-85 years
* Able to walk independently 10 meters without any gait aid (for example: walker, cane);

Exclusion Criteria:

* Unable to understand English;
* Parkinsonism or any neurological disorder with residual motor deficit (e.g.: stroke, epilepsy);
* Musculoskeletal disorder detected by clinical examination which affects gait performance;
* Active osteoarthritis affecting the lower limbs at clinical evaluation
* Use of psychotropics which can affect motor performance (e.g. neuroleptics and benzodiazepines)
* Severe Depression (score > 12/15 on the Geriatric Depression Scale).

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants 60 years or older are being recruited from the community, our Geriatrics and Memory Clinics at University of Western Ontario affiliated hospitals, from advertisements placed in local (London, ON) newspapers, and referrals from family physicians or community partners. Participants are being followed-up for up to 25 years after baseline measurements (twice annual or annual follow-up visits).
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2007-12; Primary Completion 2033-01 (Estimated); Study Completion 2033-01 (Estimated)

PRIMARY OUTCOMES:
Progression to Dementia | 25 years of follow-up
  The primary outcome is "progression to dementia" ascertained by clinician investigator using DSM-IV-TR (from 2007 to 2013) and DSM V (from 2014 and onwards). At the time of diagnosis, clinicians are blinded to baseline gait or baseline neuro-psychological test scores. Participants are being re-assessed after six months of the time point of ascertainment of dementia to confirm dementia status.
Type of Dementia | 25 years of follow-up
  Type of dementia is being established using standardized criteria for Alzheimer's disease (AD) dementia, frontotemporal dementia, Lewy body dementia, and vascular dementia (VaD).

SECONDARY OUTCOMES:
Development of Mobility Decline | 25 years of follow-up
  It is expected that MCI individuals with higher gait variability at baseline will develop mobility decline, defined as incident slowing in gait velocity (cm/s) by 10 cm/s
Incidence of Falls | 25 years of follow-up
  Falls is defined as 'an unintentionally coming to rest on the ground, floor, or other lower level and not due to a seizure or an acute stroke. Recurrent falls are defined as two or more events in a 12 months period. This outcome will be analyzed as the rate of falls over 36 months (defined as number of falls person-time at risk), the proportion of participants who fall (0, 1) and the proportion of recurrent fallers (2+ falls).
Brain anatomical changes (grey matter) | 25 years of follow-up
  Changes in grey matter volume are being as absolute change (in cm3) across assessments
Brain anatomical changes (white matter) | 25 years of follow-up
  Changes in white matter volume is being evaluated as absolute change (in cm3) across assessments.
Brain anatomical changes (ventricular volume) | 25 years of follow-up
  Changes in ventricular volume is being evaluated as absolute change (in cm3) across assessments
Mortality | 25 years of follow up
  When a participant pass away informed/documented by caregiver or medical record

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Manuel Montero Odasso, M.D., Principal Investigator — Director, Gait and Brain Lab
Locations (1):
- Gait and Brain Lab, Parkwood Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pieruccini-Faria F, Sarquis-Adamson Y, Montero-Odasso M. Mild Cognitive Impairment Affects Obstacle Negotiation in Older Adults: Results from "Gait and Brain Study". Gerontology. 2019;65(2):164-173. doi: 10.1159/000492931. Epub 2018 Oct 12. PMID 30317237
- [Background] Pieruccini-Faria F, Muir-Hunter SW, Montero-Odasso M. Do depressive symptoms affect balance in older adults with mild cognitive impairment? Results from the "gait and brain study". Exp Gerontol. 2018 Jul 15;108:106-111. doi: 10.1016/j.exger.2018.04.004. Epub 2018 Apr 10. PMID 29653157
- [Background] Montero-Odasso M, Speechley M, Muir-Hunter SW, Sarquis-Adamson Y, Sposato LA, Hachinski V, Borrie M, Wells J, Black A, Sejdic E, Bherer L, Chertkow H; Canadian Gait and Cognition Network. Motor and Cognitive Trajectories Before Dementia: Results from Gait and Brain Study. J Am Geriatr Soc. 2018 Sep;66(9):1676-1683. doi: 10.1111/jgs.15341. Epub 2018 Apr 2. PMID 29608780
- [Background] Montero-Odasso M, Speechley M. Falls in Cognitively Impaired Older Adults: Implications for Risk Assessment And Prevention. J Am Geriatr Soc. 2018 Feb;66(2):367-375. doi: 10.1111/jgs.15219. Epub 2018 Jan 10. PMID 29318592
- [Background] Montero-Odasso M, Camicioli R, Muir-Hunter SW. Dual-Task Gait And Incident Dementia-A Step Forward, But Not There Yet-Reply. JAMA Neurol. 2017 Nov 1;74(11):1380-1381. doi: 10.1001/jamaneurol.2017.2880. No abstract available. PMID 29049479
- [Background] Sakurai R, Montero-Odasso M. Apolipoprotein E4 Allele and Gait Performance in Mild Cognitive Impairment: Results From the Gait and Brain Study. J Gerontol A Biol Sci Med Sci. 2017 Nov 9;72(12):1676-1682. doi: 10.1093/gerona/glx075. PMID 28482102
- [Background] Montero-Odasso MM, Barnes B, Speechley M, Muir Hunter SW, Doherty TJ, Duque G, Gopaul K, Sposato LA, Casas-Herrero A, Borrie MJ, Camicioli R, Wells JL. Disentangling Cognitive-Frailty: Results From the Gait and Brain Study. J Gerontol A Biol Sci Med Sci. 2016 Nov;71(11):1476-1482. doi: 10.1093/gerona/glw044. Epub 2016 Mar 16. PMID 26984391
- [Background] Montero-Odasso M, Sarquis-Adamson Y, Song HY, Bray NW, Pieruccini-Faria F, Speechley M. Polypharmacy, Gait Performance, and Falls in Community-Dwelling Older Adults. Results from the Gait and Brain Study. J Am Geriatr Soc. 2019 Jun;67(6):1182-1188. doi: 10.1111/jgs.15774. Epub 2019 Jan 30. PMID 30698285
- [Background] Pieruccini-Faria F, Montero-Odasso M. Obstacle Negotiation, Gait Variability, and Risk of Falling: Results From the "Gait and Brain Study". J Gerontol A Biol Sci Med Sci. 2019 Aug 16;74(9):1422-1428. doi: 10.1093/gerona/gly254. PMID 30380013
- [Background] Pieruccini-Faria F, Hassan Haddad SM, Bray NW, Sarquis-Adamson Y, Bartha R, Montero-Odasso M. Brain Structural Correlates of Obstacle Negotiation in Mild Cognitive Impairment: Results from the Gait and Brain Study. Gerontology. 2023;69(9):1115-1127. doi: 10.1159/000530796. Epub 2023 Apr 25. PMID 37166343
- [Background] Pieruccini-Faria F, Black SE, Masellis M, Smith EE, Almeida QJ, Li KZH, Bherer L, Camicioli R, Montero-Odasso M. Gait variability across neurodegenerative and cognitive disorders: Results from the Canadian Consortium of Neurodegeneration in Aging (CCNA) and the Gait and Brain Study. Alzheimers Dement. 2021 Aug;17(8):1317-1328. doi: 10.1002/alz.12298. Epub 2021 Feb 16. PMID 33590967
- [Background] Montero-Odasso M, Oteng-Amoako A, Speechley M, Gopaul K, Beauchet O, Annweiler C, Muir-Hunter SW. The motor signature of mild cognitive impairment: results from the gait and brain study. J Gerontol A Biol Sci Med Sci. 2014 Nov;69(11):1415-21. doi: 10.1093/gerona/glu155. Epub 2014 Sep 2. PMID 25182601
- [Background] Osman A, Speechley M, Ali S, Montero-Odasso M. Fall-Risk-Increasing Drugs and Gait Performance in Community-Dwelling Older Adults: Exploratory Results from the Gait and Brain Study. Drugs Aging. 2023 Aug;40(8):721-730. doi: 10.1007/s40266-023-01045-1. Epub 2023 Jun 22. PMID 37347412
- [Background] Sakurai R, Bartha R, Montero-Odasso M. Entorhinal Cortex Volume Is Associated With Dual-Task Gait Cost Among Older Adults With MCI: Results From the Gait and Brain Study. J Gerontol A Biol Sci Med Sci. 2019 Apr 23;74(5):698-704. doi: 10.1093/gerona/gly084. PMID 29767690
- [Background] Montero-Odasso MM, Sarquis-Adamson Y, Speechley M, Borrie MJ, Hachinski VC, Wells J, Riccio PM, Schapira M, Sejdic E, Camicioli RM, Bartha R, McIlroy WE, Muir-Hunter S. Association of Dual-Task Gait With Incident Dementia in Mild Cognitive Impairment: Results From the Gait and Brain Study. JAMA Neurol. 2017 Jul 1;74(7):857-865. doi: 10.1001/jamaneurol.2017.0643. PMID 28505243
- [Background] Snir JA, Bartha R, Montero-Odasso M. White matter integrity is associated with gait impairment and falls in mild cognitive impairment. Results from the gait and brain study. Neuroimage Clin. 2019;24:101975. doi: 10.1016/j.nicl.2019.101975. Epub 2019 Aug 6. PMID 31421507
- [Background] Montero-Odasso M, Annweiler C, Hachinski V, Islam A, Yang N, Vasudev A. Vascular burden predicts gait, mood, and executive function disturbances in older adults with mild cognitive impairment: results from the gait and brain study. J Am Geriatr Soc. 2012 Oct;60(10):1988-90. doi: 10.1111/j.1532-5415.2012.04180.x. No abstract available. PMID 23057459
- [Background] Annweiler C, Beauchet O, Bartha R, Montero-Odasso M; WALK Team-Working group Angers-London for Knowledge. Slow gait in MCI is associated with ventricular enlargement: results from the Gait and Brain Study. J Neural Transm (Vienna). 2013 Jul;120(7):1083-92. doi: 10.1007/s00702-012-0926-4. Epub 2012 Nov 30. PMID 23196981
- [Background] Figgins E, Choi YH, Speechley M, Montero-Odasso M. Associations Between Potentially Modifiable and Nonmodifiable Risk Factors and Gait Speed in Middle- and Older-Aged Adults: Results From the Canadian Longitudinal Study on Aging. J Gerontol A Biol Sci Med Sci. 2021 Sep 13;76(10):e253-e263. doi: 10.1093/gerona/glab008. PMID 33420785